CLINICAL TRIAL: NCT04259892
Title: Viral Excretion in Contact Subjects at High/Moderate Risk of Coronavirus 2019-nCoV Infection
Brief Title: Viral Excretion in Contact Subjects at High/Moderate Risk of Coronavirus 2019-nCoV Infection. COVID-19.
Acronym: Cov-CONTACT
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-06; 2020-A00280-39 (Registry Identifier: RCB ID)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Coronavirus
Keywords: contact subject; high/moderate risk of transmission
MeSH Terms: conditions — Coronavirus Infections | interventions — 2019-novel coronavirus real-time reverse transcriptase diagnostic panel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: 2019-nCoV PCR — Nasopharyngeal swabs

SUMMARY:
In December 2019, a pneumonia due to a novel coronavirus (SARS-CoV-2) emerged in the city of Wuhan, in China. In a few weeks, the number of confirmed cases of SARS-CoV-2 infection has dramatically increased, with almost 150'000 cases and more than 6'000 reported deaths on March, 16th 2020.

Little is known on the rate of human-to-human transmission of this new coronavirus SARS-CoV-2 in the community and within the hospital.

Depending on the country, contact subjects considered to be at high or moderate risk of SARS-CoV-2 are, either isolated at home for a period of time defined by the health authorities or, on the contrary, continue their professional activity on the condition that they adopt measures to prevent transmission to those around them. In most European countries, healthcare workers adopt this second option. In all cases, it is most often recommended that contact persons monitor their state of health and communicate it to the persons dedicated to this action.

Whether such subjects become spreaders of the virus is not known, nor is the proportion of viral spreader who will develop a symptomatic infection.

DETAILED DESCRIPTION:
Procedures added by the research:

Phone calls for collection of reported symptoms. Nasopharyngeal swabs for determination of the presence of SARS-CoV-2 detected by PCR.

Blood sampling for determination of the presence of SARS-CoV-2 IgM or IgG. Saliva or blood sampling for whole exome sequencing of the subject.

ELIGIBILITY:
Inclusion Criteria:

1. High/moderate risk contact with a laboratory-confirmed SARS-CoV-2 case;
2. Within the 14 days following the last contact with a laboratory-confirmed SARS-CoV-2 case;
3. Obtaining informed consent.

Exclusion Criteria:

* Subject deprived of freedom
* Subject under a legal protective measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is represented by all subjects who had a contact with laboratory-confirmed SARS-CoV-2 cases and whose contact was considered to be at high/moderate risk of SARS-CoV-2 acquisition.
  This include both children and adult subjects, and healthcare workers. It may also include subject without social security in some countries, according to local legislation.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Time to SARS-CoV-2 nasopharyngeal excretion, from the day of the first high/moderate risk contact to 12 days after the last high/moderate risk contact with a laboratory-confirmed SARS-CoV-2 case. | 12 days (+/-2)
  PCR at day 0, day 3, day 5, day 7 and day 12 following the last high/moderate risk contact

SECONDARY OUTCOMES:
Time to apparition of any symptom suggestive of SARS-CoV-2 from the day of the first high/moderate risk contact to 12 days after the last high/moderate risk contact with a laboratory-confirmed SARS-CoV-2 case. | 12 days (+/-2)
  Patient Reported Outcome assessed daily (fever > 38°C, asthenia/fatigue/malaise, headache, thrills/sweating, myalgia/aches, cough, dyspnea, Acute Respiratory Distress Syndrome, diarrhea, abdominal pain, ...)
Factors associated with the time to SARS-CoV-2 nasopharyngeal excretion | 12 days (+/-2)
  nasopharyngeal excretion assessed by PCR at day 0, day 3, day 5, day 7 and day 12 following the last high/moderate risk contact
Factors associated with the time to apparition of any symptom suggestive of SARS-CoV-2 infection | 12 days (+/-2)
  Patient Reported Outcome assessed daily (fever > 38°C, asthenia/fatigue/malaise, headache, thrills/sweating, myalgia/aches, cough, dyspnea, Acute Respiratory Distress Syndrome, diarrhea, abdominal pain, ...)
Proportion of contact subjects with apparition of any symptom suggestive of SARS-CoV-2 infection | 12 days (+/-2)
  Patient Reported Outcome assessed daily (fever > 38°C, asthenia/fatigue/malaise, headache, thrills/sweating, myalgia/aches, cough, dyspnea, Acute Respiratory Distress Syndrome, diarrhea, abdominal pain, ...)
Proportion of contact subjects with positive serology defined as the presence of SARS-CoV-2 IgM or IgG at day 30 (+/-7) following last contact | 30 days (+/-7)
  ELISA, microneutralisation essay
Host genetic variants | 1 day
  Whole exome sequencing
The time (days) between the first positive SARS-CoV-2 serology and the first negative SARS-CoV-2 serology. | 365 days (+/-30)
  ELISA, microneutralisation essay

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (16):
- France (15):
  - Service de maladies infectieuses et tropicales Hôpital Jean Minjoz CHRU Besançon, Besançon
  - Service des Maladies infectieuses et tropicales, Pôle Spécialités médicales, CHU Pellegrin, Bordeaux
  - Service des maladies infectieuses Hôpital Gabriel Montpied CHU de Clermont Ferrand, Clermont-Ferrand
  - Centre d'investigation clinique 1432 Hôpital François Mitterrand CHU Bourgogne, Dijon
  - Centre d'investigation clinique 1406 CHU Grenoble, Grenoble
  - Centre d'Investigation Clinique 1403 -CHU Lille, Lille
  - Centre Investigation Clinique 1433 CHRU de NANCY, Nancy
  - Centre d'Investigation Clinique Hôpital Saint Louis, Paris
  - Centre d'investigation Clinique 1425, Hôpital Bichat Claude Bernard, Paris
  - Centre Investigation Clinique 1417 Hôpital Cochin Bâtiment Lavoisier, Paris
  - Centre d'investigation clinique 1414 Service de Pharmacologie clinique CHU Rennes Hôpital Pontchaillou, Rennes
  - Centre Hospitalier Félix Guyon Ile de la Réunion CHU nord, Saint-Denis
  - Département maladie infectieux CHU Saint Etienne, Saint-Etienne
  - Centre d'Investigation Clinique Ile de la Réunion CHU sud, Saint-Pierre
  - Centre Investigation Clinique 1415 CHRU Tours - Hôpital Bretonneau, Tours
- Service de Maladies infectieuses et tropicales Centre hospitalier, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Matuozzo D, Talouarn E, Marchal A, Zhang P, Manry J, Seeleuthner Y, Zhang Y, Bolze A, Chaldebas M, Milisavljevic B, Gervais A, Bastard P, Asano T, Bizien L, Barzaghi F, Abolhassani H, Abou Tayoun A, Aiuti A, Alavi Darazam I, Allende LM, Alonso-Arias R, Arias AA, Aytekin G, Bergman P, Bondesan S, Bryceson YT, Bustos IG, Cabrera-Marante O, Carcel S, Carrera P, Casari G, Chaibi K, Colobran R, Condino-Neto A, Covill LE, Delmonte OM, El Zein L, Flores C, Gregersen PK, Gut M, Haerynck F, Halwani R, Hancerli S, Hammarstrom L, Hatipoglu N, Karbuz A, Keles S, Kyheng C, Leon-Lopez R, Franco JL, Mansouri D, Martinez-Picado J, Metin Akcan O, Migeotte I, Morange PE, Morelle G, Martin-Nalda A, Novelli G, Novelli A, Ozcelik T, Palabiyik F, Pan-Hammarstrom Q, de Diego RP, Planas-Serra L, Pleguezuelo DE, Prando C, Pujol A, Reyes LF, Riviere JG, Rodriguez-Gallego C, Rojas J, Rovere-Querini P, Schluter A, Shahrooei M, Sobh A, Soler-Palacin P, Tandjaoui-Lambiotte Y, Tipu I, Tresoldi C, Troya J, van de Beek D, Zatz M, Zawadzki P, Al-Muhsen SZ, Alosaimi MF, Alsohime FM, Baris-Feldman H, Butte MJ, Constantinescu SN, Cooper MA, Dalgard CL, Fellay J, Heath JR, Lau YL, Lifton RP, Maniatis T, Mogensen TH, von Bernuth H, Lermine A, Vidaud M, Boland A, Deleuze JF, Nussbaum R, Kahn-Kirby A, Mentre F, Tubiana S, Gorochov G, Tubach F, Hausfater P; COVID Human Genetic Effort; COVIDeF Study Group; French COVID Cohort Study Group; CoV-Contact Cohort; COVID-STORM Clinicians; COVID Clinicians; Orchestra Working Group; Amsterdam UMC Covid-19 Biobank; NIAID-USUHS COVID Study Group; Meyts I, Zhang SY, Puel A, Notarangelo LD, Boisson-Dupuis S, Su HC, Boisson B, Jouanguy E, Casanova JL, Zhang Q, Abel L, Cobat A. Rare predicted loss-of-function variants of type I IFN immunity genes are associated with life-threatening COVID-19. Genome Med. 2023 Apr 5;15(1):22. doi: 10.1186/s13073-023-01173-8. PMID 37020259